CLINICAL TRIAL: NCT06605508
Title: Prospective Observational Study on Intracavernosal Injection of Autologous Adipose Tissue-Derived Stem Cells (ADSC) or Stem Cell-derived Exosomes for the Treatment of Erectile Dysfunction
Brief Title: Regenerative Injection of Stem Cells or Stem Cell-derived Exosomes for Erectile Dysfunction (RISE)
Acronym: RISE
Status: Recruiting | Type: Observational
Sponsor: Jumeirah American Clinic (Other)
Responsible Party: Principal Investigator, Ranjith Ramasamy, Consultant Urologist, Jumeirah American Clinic
Other Study IDs: 001
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Associated With Type 2 Diabetes Mellitus; Erectile Dysfunction Following Radical Prostatectomy
Keywords: stem cell therapy; Erectile dysfunction (ED); Autologous adipose tissue-derived stem cells (ADSC); Regenerative medicine for ED; Exosomes
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intracavernosal Injection of Autologous Adipose Stem Cells for Erectile Dysfunction Treatment: In this arm of the study, participants will receive intracavernosal injections of autologous adipose tissue-derived stem cells (ADSC). The ADSC are collected from the participant's own body fat through a minimally invasive liposuction procedure. After processing, the stem cells will be injected directly into the erectile tissue of the penis. This treatment aims to improve erectile function by stimulating tissue regeneration and enhancing blood flow. Participants will be monitored for safety and efficacy, including erectile function assessments using the International Index of Erectile Function (IIEF) and penile hemodynamics measured by Doppler ultrasound. Follow-up evaluations will occur at 3, 6, 9, and 12 months post-treatment.
  Interventions: Procedure: Autologous Adipose Tissue-Derived Stem Cell Injection for Erectile Dysfunction
- Intracavernosal Injection of Stem cell-derived exosomes: In this arm of the study, participants will receive intracavernosal injections of stem cell-derived exosomes. These exosomes, which are nano-sized extracellular vesicles obtained from cultured stem cells, are rich in growth factors and bioactive molecules that facilitate tissue repair and regeneration. Unlike stem cell therapy, this cell-free approach minimizes potential risks associated with live cell transplantation while still delivering therapeutic benefits. Participants will be monitored for safety and efficacy, including erectile function assessments using the International Index of Erectile Function (IIEF) and penile hemodynamics measured by Doppler ultrasound. Follow-up evaluations will occur at 3, 6, 9, and 12 months post-treatment.
  Interventions: Procedure: Stem cell-derived Exosomes Injection for Erectile Dysfunction

INTERVENTIONS:
Procedure: Autologous Adipose Tissue-Derived Stem Cell Injection for Erectile Dysfunction — This intervention involves the use of autologous adipose tissue-derived stem cells (ADSC) to treat erectile dysfunction. The process begins with a minimally invasive liposuction procedure to harvest fat tissue from the participant's own body. The harvested fat is then processed to isolate stem cells, which are subsequently injected directly into the erectile tissue of the penis. This approach aims to enhance erectile function by promoting tissue regeneration and improving blood flow. Unlike other treatments for erectile dysfunction, this intervention uses stem cells derived from the participant's own fat, which may reduce the risk of immune rejection and offer a novel regenerative therapy option. The treatment is designed to address ED in patients who have not responded adequately to conventional therapies like PDE-5 inhibitors.
  Other Names: ADSC Injection for ED; Fat-Derived Stem Cell Therapy for Erectile Dysfunction; Autologous Fat Stem Cell Injection
  Groups: Intracavernosal Injection of Autologous Adipose Stem Cells for Erectile Dysfunction Treatment
Procedure: Stem cell-derived Exosomes Injection for Erectile Dysfunction — This intervention involves the use of stem cell-derived exosomes to treat erectile dysfunction. Exosomes are nano-sized extracellular vesicles secreted by stem cells, containing bioactive molecules such as growth factors and signaling proteins that promote tissue repair and regeneration. Unlike therapies requiring the transplantation of live cells, this cell-free approach eliminates the need for invasive harvesting procedures. The exosomes are carefully purified from cultured stem cells and prepared for direct injection into the erectile tissue of the penis. This approach aims to enhance erectile function by stimulating tissue regeneration, reducing inflammation, and improving blood flow. Unlike other treatments for erectile dysfunction, exosome therapy offers a novel regenerative option, potentially benefiting patients who have not responded adequately to conventional therapies such as PDE-5 inhibitors.
  Other Names: Extracellular Vesicle Therapy; Cell-Free Regenerative Therapy for ED
  Groups: Intracavernosal Injection of Stem cell-derived exosomes

SUMMARY:
The goal of this prospective observational study is to evaluate whether injections of stem cells derived from the patient's own fat tissue (adipose tissue) can improve erectile function in men aged 30 to 75 who have erectile dysfunction (ED) and have not responded well to standard treatments like PDE-5 inhibitors (e.g., Viagra).

The main questions the study aims to answer are:

Will the stem cell injections improve erectile function, as measured by the International Index of Erectile Function (IIEF) score? Are there any changes in blood flow to the penis, which will be measured using a Doppler ultrasound?

Participants will:

Receive injections of their own stem cells (obtained from a biopsy of fat) directly into the penis.

Undergo assessments to check erectile function before and after treatment. Have follow-up visits at 3, 6, 9, and 12 months to monitor long-term effects. The study will also look for any possible side effects or complications and evaluate biological markers in the penis that may indicate the effectiveness of the treatment.

Participants will be recruited from clinic where they are already receiving care for ED. To take part, they must be in good overall health, with no severe heart disease, uncontrolled diabetes, cancer, or other conditions that could make stem cell therapy unsafe for them.

DETAILED DESCRIPTION:
Detailed Description:

This prospective observational study is designed to evaluate the safety and preliminary efficacy of intracavernosal injections of autologous adipose tissue-derived stem cells (ADSCs) or stem cell-derived exosomes for treating erectile dysfunction (ED) in men unresponsive to conventional therapies, such as phosphodiesterase type 5 (PDE-5) inhibitors. The primary focus will be on improvements in erectile function, as measured by changes in the International Index of Erectile Function (IIEF) score. Additionally, the study will assess penile hemodynamics, monitor adverse events, and explore biomarkers that may predict therapeutic outcomes.

Background and Rationale:

Erectile dysfunction affects a significant proportion of the male population, particularly with advancing age, and can result from various causes, including vascular, neurogenic, and psychogenic factors. Current standard treatments, such as PDE-5 inhibitors, are effective for many, but a substantial subset of patients-especially those with underlying vascular or nerve-related pathologies-experience inadequate therapeutic responses.

Regenerative medicine has emerged as a promising approach for addressing ED through tissue repair and vascular regeneration. Both ADSCs and stem cell-derived exosomes are potential therapies due to their ability to promote angiogenesis, tissue regeneration, and anti-inflammatory effects. ADSCs can be harvested from the patient's adipose tissue, minimizing the risk of immunogenicity or rejection. Exosomes derived from stem cells, on the other hand, offer a cell-free approach, delivering growth factors and signaling molecules to the target tissues. Preclinical studies have demonstrated the potential of these therapies to restore erectile function through tissue remodeling and enhanced penile blood flow following intracavernosal injection.

Primary Objective:

To evaluate the safety and efficacy of intracavernosal ADSC or stem cell-derived exosome injections in improving erectile function, as determined by changes in the IIEF score from baseline through subsequent follow-ups. The IIEF is a validated, comprehensive questionnaire used to assess erectile function and sexual satisfaction.

Secondary Objectives:

Penile Hemodynamics: Doppler ultrasound will evaluate changes in penile blood flow post-treatment, providing insight into the vascular effects of the therapies.

Long-Term Effects: Follow-up visits at 3, 6, 9, and 12 months will include IIEF scoring, Doppler ultrasound assessments, and patient-reported outcomes to evaluate the durability of treatment effects.

Safety and Adverse Events: All potential adverse events, including injection-site reactions and systemic complications, will be closely monitored and documented throughout the study.

Biomarker Exploration: Exploratory analyses will aim to identify biomarkers, including vascular and tissue-specific markers, which may predict patient response to the treatment.

Study Design:

This open-label, single-arm, pilot observational study will serve as a preliminary investigation of ADSC or stem cell-derived exosome therapy in ED, providing foundational data on their feasibility and safety. As a prospective observational study, the emphasis will be on safety and gathering initial efficacy data rather than delivering definitive conclusions.

Study Population:

The study will enroll 30 men aged 30 to 75 years with a diagnosis of mild to moderate erectile dysfunction who have failed or experienced suboptimal responses to PDE-5 inhibitors. Participants will be recruited from Dr. Ranjith Ramasamy's clinic, where they are receiving care for ED. Inclusion and exclusion criteria have been carefully designed to select participants who are most likely to benefit from these therapies and ensure patient safety.

Sample Size Rationale:

A sample size of 30 was chosen based on the exploratory nature of the study. The primary goal is to assess feasibility, safety, and preliminary efficacy while providing sufficient data to inform the design of future, more extensive studies. Recruitment of 30 participants is feasible within the clinic's patient population over the planned two-year period.

Study Procedures:

Informed Consent: Participants will be fully informed about the study, including its risks and benefits, and will provide written consent prior to enrollment.

Baseline Assessments: Baseline data, including IIEF scores, penile Doppler ultrasound, and blood tests, will be collected to assess pre-treatment erectile function and overall health.

Therapeutic Administration:

For ADSCs: ADSCs will be isolated from autologous adipose tissue harvested via minimally invasive liposuction. The cells will be processed and prepared for direct injection into the corpus cavernosum. A tourniquet will be placed for 15 minutes around the base of the penis after the injection to minimize systemic dispersion.

For Exosomes: Exosomes derived from stem cells will be isolated and purified, then injected intracavernosally using a similar protocol.

Follow-Up Monitoring: Participants will be monitored for immediate post-injection reactions and at regular intervals (3, 6, 9, and 12 months) for changes in erectile function (IIEF), penile hemodynamics (Doppler ultrasound), and adverse events. Exploratory biomarker analysis will also be conducted.

Data Collection and Analysis:

Data will be analyzed to evaluate primary and secondary outcomes. IIEF score changes will be the primary efficacy measure, while penile hemodynamics and adverse event rates will be assessed for safety. Exploratory analyses will investigate the correlation between biomarkers and clinical outcomes, providing insights into potential predictors of treatment response.

Ethical Considerations:

This study will adhere to ethical standards for clinical research. Informed consent will be obtained from all participants, and the protocol will be reviewed and approved by an ethics committee. Participants will have the right to withdraw at any point, and their standard medical care will not be affected by their participation.

Expected Outcomes:

The study aims to provide early evidence on the safety and potential efficacy of ADSC or stem cell-derived exosome therapy for ED. If successful, participants are expected to show improvements in erectile function with minimal adverse events. The findings from this study will inform larger, more definitive trials and contribute to the development of novel regenerative therapies for erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adult males aged 30 to 75 years.
* Diagnosis: Confirmed diagnosis of erectile dysfunction (ED) of mild to moderate severity, as defined by an International Index of Erectile Function (IIEF) score.
* Treatment Response: Failure or suboptimal response to conventional ED treatments, such as PDE-5 inhibitors.
* General Health: Overall good health without contraindications to stem cell therapy.
* Informed Consent: Ability and willingness to provide written informed consent to participate in the study.

Exclusion Criteria:

* Severe Cardiovascular Disease: Presence of severe cardiovascular conditions, including uncontrolled hypertension or significant heart disease.
* Active Infections: Ongoing infections that could interfere with treatment or pose a risk to the participant.
* Malignancies: History of or current cancer, including malignancies that could affect safety or treatment outcomes.
* Contraindications to Stem Cell Therapy: Any medical conditions or treatments that contraindicate the use of stem cell therapy.
* Uncontrolled Diabetes: Poorly controlled diabetes or other metabolic disorders that could impact treatment efficacy or safety.
* Psychiatric or Cognitive Impairments: Significant psychiatric or cognitive disorders that may affect the participant's ability to comply with study protocols or provide informed consent.
* Recent Surgery or Trauma: Recent major surgeries or physical trauma that could impact the study or interfere with the intervention.
* Participation in Other Studies: Participation in other clinical trials or studies that may affect the outcomes or safety of this study.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of men aged 30 to 75 years with a clinical diagnosis of mild to moderate erectile dysfunction (ED). Eligible participants are those who have experienced suboptimal or no response to standard therapies, including phosphodiesterase type 5 (PDE-5) inhibitors. The inclusion criteria are designed to focus on individuals most likely to benefit from regenerative therapy while ensuring safety.
  Participants will be recruited from Dr. Ranjith Ramasamy's clinic, where they are actively seeking care for erectile dysfunction. This population is expected to represent a diverse group of patients with varying etiologies of ED, including vascular, neurogenic, and idiopathic causes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Erectile Function as Measured by the International Index of Erectile Function (IIEF) Score | 12 months
  The primary outcome measure for this study is the change in erectile function as assessed by the International Index of Erectile Function (IIEF) score. The IIEF is a validated questionnaire designed to evaluate various aspects of sexual health, including erectile function, sexual satisfaction, and overall sexual performance. Participants will complete the IIEF questionnaire at baseline and at follow-up visits to track changes in erectile function over time. The goal is to determine whether the intracavernosal injection of autologous adipose tissue-derived stem cells leads to significant improvements in erectile function compared to pre-treatment levels. The IIEF score will provide a comprehensive measure of treatment effectiveness and help assess the impact of the intervention on participants' sexual health and quality of life.

SECONDARY OUTCOMES:
Penile Hemodynamics as Measured by Doppler Ultrasound | 12 months
  The secondary outcome measure for this study is penile hemodynamics assessed by Doppler ultrasound. Doppler ultrasound is a non-invasive imaging technique used to evaluate blood flow and vascular function in the penis. This assessment will be conducted at baseline and during follow-up visits to determine changes in penile blood flow and vascular characteristics following the intracavernosal injection of autologous adipose tissue-derived stem cells. Improvements in penile hemodynamics, such as increased blood flow and better vascular function, will be used to gauge the effectiveness of the stem cell therapy in enhancing erectile function. This measure will complement changes in the International Index of Erectile Function (IIEF) score and provide a detailed understanding of the physiological effects of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Jumeirah American Clinic, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, gender, and relevant medical history. Baseline Assessments: Initial International Index of Erectile Function (IIEF) scores, Doppler ultrasound measurements, and other relevant baseline data.
  Treatment Data: Details of the autologous adipose tissue-derived stem cell injections, including dosage and administration specifics.
  Follow-Up Data: Changes in IIEF scores and Doppler ultrasound measurements at follow-up points (3, 6, 9, and 12 months).
  Adverse Events: Documentation of any adverse events or complications experienced during the study.
Supporting Information: Study Protocol, ICF
Time Frame: January 1, 2025 to December 31, 2027
Access Criteria: Access to individual participant data (IPD) and supporting information from this study will be managed according to the following criteria:
  Eligible Users: Access will be granted to qualified researchers, academic institutions, and regulatory bodies who have a legitimate interest in the data, such as those conducting further analyses or validating study findings.
  Data Access:
  Research Data: Includes de-identified demographic information, baseline assessments, treatment data, follow-up results, adverse event reports, and biomarker data.
  Supporting Information: Includes study protocols, informed consent forms, and other relevant documentation.
  Access Process:
  Request Submission: Interested parties must submit a formal request detailing the purpose of data use and how the data will be used.
  Review and Approval: Requests will be reviewed by the study's data access committee or a designated review board to ensure they meet ethical and scientific standards.

REFERENCES:
- [Background] Narasimman M, Sandler M, Bernstein A, Loloi J, Saltzman RG, Bernie H, Ramasamy R. A primer on the restorative therapies for erectile dysfunction: a narrative review. Sex Med Rev. 2024 Jun 26;12(3):505-512. doi: 10.1093/sxmrev/qeae012. PMID 38494449